CLINICAL TRIAL: NCT00135993
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Five-Arm Parallel-Group Trial to Investigate the Efficacy and Safety of Four Different Transdermal Doses of Rotigotine in Subjects With Idiopathic Restless Legs Syndrome
Brief Title: Four Different Transdermal Doses of Rotigotine in Subjects With Idiopathic Restless Legs Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP0792
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Restless Legs Syndrome
Keywords: Idiopathic Restless Leg syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — rotigotine

INTERVENTIONS:
Drug: Rotigotine

SUMMARY:
Subjects who meet the diagnosis of idiopathic restless legs syndrome (RLS) based on the 4 cardinal clinical features according to the International Restless Legs Syndrome Study Group (IRLSSG) are allowed to enroll in this trial.

The primary objective of this trial is to demonstrate that rotigotine (SPM 936) is efficacious in subjects with idiopathic restless legs syndrome. Additional objectives are to investigate the safety and tolerability of rotigotine.

Subjects will be randomized to receive either placebo, 1.125, 2.25, 4.5, or 6.75mg/day rotigotine in a 1:1:1:1:1 (active:placebo) fashion. Approximately 600 subjects will be enrolled in this trial, participating at approximately 60 sites. The maximum duration of the trial is approximately 8 months (consisting of a 4-week Titration Period, a 6-month Maintenance Period, a 7-day Taper Period, and a 30-day Safety Follow-Up Period).

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic restless legs syndrome

Exclusion Criteria:

* History of sleep disturbances

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 811 (Actual)
Dates: Start 2005-05; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
IRLS sum score and CGI Item 1 score severity of illness | From Baseline at the end of the Maintenance Period

SECONDARY OUTCOMES:
IRLS Responder: A responder is a subject with a decrease of ≥50% in IRLS sum score | From Baseline at the end of the Maintenance Period
CGI Item 1 Responder: A responder is defined as a subject with a decrease of ≥50% in CGI Item 1 | From Baseline at the end of the Maintenance Period
Changes in CGI Items 2-3 (continuous) during the Maintenance Period; Change from Baseline in RLS-6 Rating Scales at the end of the Maintenance Period

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (1):
- Schwarz, RTP, North Carolina, United States

REFERENCES:
- [Result] Hening WA, Allen RP, Ondo WG, Walters AS, Winkelman JW, Becker P, Bogan R, Fry JM, Kudrow DB, Lesh KW, Fichtner A, Schollmayer E; SP792 Study Group. Rotigotine improves restless legs syndrome: a 6-month randomized, double-blind, placebo-controlled trial in the United States. Mov Disord. 2010 Aug 15;25(11):1675-83. doi: 10.1002/mds.23157. PMID 20629075
- [Derived] Ondo WG, Grieger F, Moran K, Kohnen R, Roth T. Post Hoc Analysis of Data from Two Clinical Trials Evaluating the Minimal Clinically Important Change in International Restless Legs Syndrome Sum Score in Patients with Restless Legs Syndrome (Willis-Ekbom Disease). J Clin Sleep Med. 2016 Jan;12(1):63-70. doi: 10.5664/jcsm.5396. PMID 26446245